CLINICAL TRIAL: NCT07239700
Title: Effectiveness of Buzzy and TickleFlex Applications in Reducing Pain and Fear Associated With Insulin Injections in Children With Type 1 Diabetes
Brief Title: Buzzy and TickleFlex in Reducing Insulin Injection Pain and Fear
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hakkari Universitesi (Other)
Responsible Party: Principal Investigator, Nesrullah AYŞİN, Assistant Professor, Hakkari Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HakkariU-SHMYO-NA-01
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Diabete Type 1; Diabetes in Children
Keywords: Type 1 Diabetes Mellitus; Children; Insulin Injection; Pain; Fear; Nonpharmacological Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Pain

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, parallel-assignment interventional model with three arms: Buzzy device application, TickleFlex device application, and control (standard insulin injection).
Masking Description: This study is conducted as an open-label randomized controlled trial. Due to the visible nature of the devices (Buzzy and TickleFlex), participants, parents, and the administering researcher cannot be masked to group assignments. However, outcome assessments are standardized and independently rated by three parties: the child, the parent, and the researcher, using validated pain and fear scales. This approach aims to minimize observer and reporting bias even in the absence of full blinding. No additional parties beyond those listed are masked in this clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Buzzy Device Application (Experimental): Participants received vibration and cold stimulation using the Buzzy device before and during insulin injection.
  Interventions: Device: Buzzy
- TickleFlex Device Application (Experimental): Participants used the TickleFlex device attached to their insulin pens during insulin injection.
  Interventions: Device: TickleFlex
- Standard Insulin Injection (Control) (Other): Participants received routine insulin injections without any adjunctive device or intervention.
  Interventions: Other: None (Routine Care)

INTERVENTIONS:
Device: Buzzy — The Buzzy device is a non-invasive, bee-shaped device that combines cold and vibration to reduce pain perception during needle procedures. It was applied for 30 seconds before and during insulin administration to reduce pain and fear according to the gate control theory.
  Arms: Buzzy Device Application
Device: TickleFlex — The TickleFlex device is a soft, flexible insulin-pen attachment that gently stretches the skin and diffuses needle pressure, reducing injection pain and anxiety in children with Type 1 Diabetes Mellitus.
  Arms: TickleFlex Device Application
Other: None (Routine Care) — Standard subcutaneous insulin injection performed following pediatric diabetes nursing protocols.
  Arms: Standard Insulin Injection (Control)

SUMMARY:
This interventional randomized controlled clinical trial aims to evaluate the effectiveness of two nonpharmacological devices, Buzzy and TickleFlex, in reducing pain and fear associated with insulin injections among children with Type 1 Diabetes Mellitus (T1DM).

A total of 90 participants aged 6 to 12 years will be randomly assigned to one of three groups: Buzzy, TickleFlex, or control. The Buzzy device provides combined cold and vibration stimulation near the injection site to decrease pain perception based on the gate control theory, while the TickleFlex device is a soft, flexible attachment for insulin pens designed to minimize needle pressure and discomfort during injection.

Pain and fear will be assessed immediately before and after a single insulin injection using validated instruments, including the Wong-Baker FACES Pain Rating Scale and the Children's Fear Scale (CFS), rated independently by the child, parent, and researcher.

It is hypothesized that both Buzzy and TickleFlex applications will significantly reduce pain and fear compared to standard insulin injection without intervention. The study is expected to provide evidence supporting the use of nonpharmacological methods in pediatric diabetes care to improve children's comfort and treatment adherence.

DETAILED DESCRIPTION:
Children with Type 1 Diabetes Mellitus (T1DM) require multiple daily insulin injections, which are often associated with pain, fear, and anxiety. Repeated exposure to needle-related discomfort can negatively affect children's treatment adherence, emotional well-being, and overall quality of life. Therefore, there is a growing need for safe, practical, and nonpharmacological interventions to improve the injection experience in pediatric diabetes care.

This randomized controlled trial aims to investigate the effectiveness of two noninvasive devices-Buzzy and TickleFlex-in reducing pain and fear during insulin injections in children with T1DM. The Buzzy device uses vibration and cold stimulation to reduce pain perception through the gate control mechanism, while the TickleFlex device, a soft and flexible attachment for insulin pens, minimizes needle pressure and distributes the injection sensation evenly.

A total of 90 children aged 6-12 years will be randomly assigned to three groups: Buzzy, TickleFlex, and control. All participants will receive a single subcutaneous insulin injection as part of their regular diabetes management. Pain and fear levels will be measured before and immediately after the injection using validated scales: the Wong-Baker FACES Pain Rating Scale and the Children's Fear Scale (CFS), rated independently by the child, parent, and researcher.

It is hypothesized that both Buzzy and TickleFlex will significantly reduce perceived pain and fear compared with standard insulin injection without intervention. Findings from this study are expected to contribute to evidence-based pediatric nursing practices by supporting the integration of nonpharmacological pain management methods into routine diabetes care.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 12 years.
* Diagnosed with Type 1 Diabetes Mellitus (T1DM) for at least 6 months.
* Receiving daily subcutaneous insulin injections as part of routine diabetes management.
* Able to understand and communicate pain and fear levels using the Wong-Baker -FACES Pain Rating Scale and the Children's Fear Scale.
* Accompanied by a parent or legal guardian who can provide informed consent.
* Willingness of both the child and parent to participate in the study.
* No visual, auditory, or cognitive impairments that would interfere with data collection.

Exclusion Criteria:

* Presence of neurological, sensory, or cognitive disorders that may affect pain or fear perception.
* Peripheral neuropathy or other diabetic complications influencing pain sensation.
* Use of analgesics, sedatives, or anxiolytic medications within 24 hours prior to data collection.
* Local skin lesions, infections, or allergies at or near the insulin injection site.
* History of needle phobia or severe anxiety disorders diagnosed by a healthcare professional.
* Concurrent participation in another interventional clinical study.
* Refusal or inability of the child or parent/guardian to provide written informed consent.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity During Insulin Injection | Immediately before and after a single insulin injection.
  The primary outcome is the level of pain experienced by children during insulin injection, measured using the Wong-Baker FACES Pain Rating Scale (0-10). Assessments are performed independently by the child, parent, and researcher immediately before and after the injection. Higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
Fear Level Associated with Insulin Injection | Immediately before and after a single insulin injection.
  The secondary outcome is the level of fear experienced by children during insulin injection. Fear is assessed using the Children's Fear Scale (CFS), which scores from 0 (no fear) to 4 (extreme fear). Assessments are conducted independently by the child, parent, and researcher before and immediately after the injection. Lower scores indicate reduced fear levels.

CONTACTS AND LOCATIONS:
Overall Officials: Nesrullah AYŞİN, PHD, Principal Investigator — Hakkari University
Locations (1):
- Hakkari University, Hakkâri, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available upon reasonable request to qualified researchers after publication of the primary results. Requests will be reviewed by the principal investigator to ensure compliance with ethical and data protection standards. Data will include pain and fear scores but exclude any identifiable personal information.
Supporting Information: Study Protocol, ICF
Time Frame: Not applicable. Individual participant data will not be shared.
Access Criteria: Access to de-identified individual participant data (IPD) will be available to qualified researchers who submit a reasonable written request describing the research purpose and data use plan. Requests will be evaluated by the Principal Investigator to ensure compliance with ethical standards, participant privacy, and institutional policies. Approved researchers will receive access to de-identified datasets containing pain and fear scores only, excluding any information that could directly or indirectly identify participants. Data will be shared electronically through secure, password-protected institutional channels.